CLINICAL TRIAL: NCT00026039
Title: Women's Estrogen for Stroke Trial (WEST)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Allocation: Randomized | Masking: Double
Other Study IDs: R01NS031251 (NIH)
Record Dates: First submitted 2001-11-07; First posted 2001-11-08 (Estimated); Last update posted 2006-05-15 (Estimated); Status verified 2005-11

CONDITIONS: Stroke
Keywords: stroke; estrogen
MeSH Terms: conditions — Stroke | interventions — Estrogens

INTERVENTIONS:
Drug: estrogen

SUMMARY:
To determine if estrogen hormone replacement therapy reduces the risk of stroke or death in postmenopausal women who have already had stroke or a transient ischemic attack (TIA).

DETAILED DESCRIPTION:
The researchers enrolled 664 postmenopausal women with an average age of 71 years who had experienced an ischemic stroke or a TIA within the previous 90 days. Ischemic strokes and TIAs result from blockages in the vessels that supply blood to the brain. Participants were given a number of initial assessments, including the NIH Stroke Scale (NIHSS) of neurological impairment and the Barthel index of functional ability in activities of daily living. In addition to the usual best care for patients who have had a stroke, women in the trial received either oral estrogen (estradiol 17-beta at the standard replacement dose of 1 mg daily) or a matching placebo. Patients were studied for an average of 2.8 years. They stopped receiving the estrogen or placebo if they had a stroke.

The researchers found that there was no significant difference in the incidence of stroke or death in the women who were randomly assigned to receive estrogen instead of placebo. However, they found that the incidence of death due to stroke was higher in the estrogen group and that the non-fatal strokes in that group were associated with slightly worse neurological and functional impairments at 1 month after stroke. The risk of stroke within the first 6 months after enrollment in the study was also higher among women in the estrogen group. There were no significant differences between treatment groups in the number of TIAs or non-fatal heart attacks. However, participants receiving estrogen were more likely to experience gynecologic complications, particularly vaginal bleeding.

Age Groups: Child, Adult, Older Adult
Dates: Start 1993-12

CONTACTS AND LOCATIONS:
Overall Officials: Ralph I. Horwitz, M.D., Principal Investigator — Yale University